CLINICAL TRIAL: NCT05835700
Title: Research of the Relationship Between Serum Gasdermin-d Levels and Pyroptosis and Preterm Labor
Brief Title: The Relationship Between Serum Gasdermin-D Levels and Pyroptosis and Preterm Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Nefise Nazlı YENIGUL, Ph.D. Assistant Professor Department of Obstetrics and Gynecology, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2011-KAEK-25 2021/06-11
Record Dates: First submitted 2023-04-04; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Gasdermin D Levels in Preterm Labor
Keywords: gasdermin D; preterm labor; pyroptosis
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Intervention Model Description: Gastermin D and Pentaxin 3 levels were measured in the patients participating in the study. These are not routinely checked markers. Participants were assigned prospectively to an intervention or interventions according to a protocol to evaluate the effect of the intervention(s) on preeclampsia or HELLP related outcomes. Due to this, our work is interventional.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gasdermin-D levels in preterm labor (study group) (Other): Maternal serum Gasdermin-D levels of pregnant women who were diagnosed with idiopathic preterm labor
  Interventions: Other: Gasdermin-d
- Gasdermin-D levels in healthy pregnant women (control group) (Other): Maternal serum Gasdermin-D levels of healthy pregnant women
  Interventions: Other: Gasdermin-d

INTERVENTIONS:
Other: Gasdermin-d — Maternal serum Gasdermin-D levels in preterm labor and healthy pregnant women.

SUMMARY:
In this study, the investigators aimed to investigate the relationship between Gasdermin D levels measured from the maternal serum of patients diagnosed with preterm labor and spontaneous preterm labor in pregnant women.

DETAILED DESCRIPTION:
This prospective case- control study was conducted between 15 July 2021 and 15 July 2022 at Bursa Yüksek İhtisas Training and Research Hospital. The study was conducted with pregnant women between the ages of 18-45 who were idiopathic preterm labor. Pregnant women between the ages of 18-45 who were diagnosed with preterm labor between 24-37 weeks of gestational were included. This study was conducted with 160 pregnant women who were diagnosed with idiopathic preterm labor and 167 healthy pregnant women who were in the same gestational week as these pregnant women and were not diagnosed with preterm labor. Group 1 patients diagnosed with preterm labor between 24-37 weeks( study group) (n:160), Group 2 consisted of healthy pregnant women who were not diagnosed with preterm labor between 24-37 weeks ( control group) (n: 167) . In group 1, 80 patients were diagnosed with early preterm (between 24-34 weeks ) and 80 patients with late preterm labor (34-36+6 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who were diagnosed with idiopathic preterm labor and gave birth in our hospital
* Pregnant women without vaginal infection
* Healthy pregnant women between 24-37 weeks without a diagnosis of preterm labor

Exclusion Criteria:

* Multiple pregnancies
* Pregnant women with a prediagnosis of chromosomal and congenital anomalies in the fetus
* Women with a known infective or autoimmune disease before pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 327 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
relationship between Gasdermin-D levels in preterm labor | 12 months
  the relationship between Gasdermin-D levels of patients diagnosed with preterm labor and spontaneous preterm labor in pregnant women.

CONTACTS AND LOCATIONS:
Locations (1):
- Nefise Nazlı YENIGUL, Bursa, Turkey (Türkiye)